CLINICAL TRIAL: NCT07273357
Title: Follow-Up After adjuvanT CDK4/6i Use in oldeR brEast Cancer Patients - Aspects on Geriatric Screening, Toxicities, and Quality of Life (FUTURE)
Brief Title: Aspects of Adjuvant CDK4/6 Inhibitors in Older Breast Cancer Patients - Focusing on Geriatric Screening
Acronym: FUTURE
Status: Not yet recruiting | Type: Observational
Sponsor: Region Jönköping County (Other Government)
Collaborators: Region Örebro County (Other); Region Östergötland (Other); Region Gävleborg (Other); Västra Götalandsregionen (Other); Linkoeping University (Other Government); Örebro University, Sweden (Other); Kalmar County Hospital (Other)
Responsible Party: Principal Investigator, Christine Lundgren, Principal Investigator, Region Jönköping County
Other Study IDs: EPM 2025-06207-01
Record Dates: First submitted 2025-11-14; First posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-11

CONDITIONS: Geriatric Assessment; Adjuvant Drug Therapy; Breast Cancer Early Stage Breast Cancer (Stage 1-3)
Keywords: Older patients; Geriatric screening; Adjuvant CDK4/6 inhibitors; Breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Frail and fit older (≥70 years) breast cancer patients: Older (≥70 years) patients, with early stage breast cancer, initiating adjuvant CDK4/6 inhibitors that are defined as frail or fit according to G8 and VES-13

SUMMARY:
Older breast cancer patients should not be categorically excluded from adjuvant therapies, including the recommended CDK4/6 inhibitors (CDK4/6i) administered in combination with endocrine therapy. Nevertheless, this population frequently presents with comorbidities that may increase susceptibility to treatment-related toxicities, including impacts on quality of life, which must be carefully considered when selecting therapeutic regimens. Given the limited representation of older patients in the clinical trials behind the recommendations for adjuvant CDK4/6i therapy, coupled with the uncertain magnitude of clinical benefit and the reported rates of toxicity and treatment discontinuation, it is essential to critically evaluate both efficacy and safety in this specific patient subgroup. National and international guidelines recommend the integration of geriatric assessments into routine clinical practice to facilitate individualized treatment decisions; however, such assessments are not yet widely implemented in many oncology departments and are not routinely in use to guide adjuvant CDK4/6i therapy.

This study aims to investigate the implementation of geriatric assessments in older breast cancer patients (≥70 years) and to examine multiple dimensions of CDK4/6i treatment in this cohort, including short- and medium-term effects on quality of life, dose intensity, and clinical outcomes. By doing so, the investigators seek to more accurately delineate the benefits and risks of adjuvant CDK4/6i therapy in this specific patient population.

DETAILED DESCRIPTION:
Adjuvant systemic therapy for breast cancer incorporates many different treatment modalities. CDK4/6 inhibitors (CDK4/6i) were initially approved in the metastatic setting, but now also as adjuvant treatment, concomitant with endocrine therapy for patients with estrogen-receptor positive/human epidermal growth factor receptor 2 -negative (ER+/HER2-) disease.

Only 15% of the study population in MonarchE was aged 65 and older, and the median age of 51 years is a decade younger than in the advanced setting pivotal studies. The median age in NATALEE was similarly 52 years, including only 773 out of 5,101 aged ≥65 years. Subgroup analysis from the MonarchE trial suggests benefit also in those >65 years old, but no statistically significant results exist so far. This might be attributed to a relatively small number of older participants, and the fact that these subgroup analyses were not pre-planned.

At present, specific guidelines regarding the use of adjuvant CDK4/6i in older patients are lacking. Given the importance of tailoring adjuvant treatment in this population, the implementation of geriatric screening in patients ≥70 years who are candidates for adjuvant CDK4/6i therapy is warranted. Furthermore, it is of clinical relevance to investigate the associations between geriatric screening assessment, quality of life, treatment-related toxicity, and discontinuation in this cohort. Outcomes such as hospitalization rates, recurrence, survival, and treatment dose intensity are also of particular interest in this patient population.

The hypothesis that the use of geriatric screening in routine clinical practice will reveal a relationship between frailty and decreased quality of life and higher risk of developing CDK4/6i toxicity. The investigators moreover anticipate a correlation between higher frailty and lower dose intensity, and poorer outcomes in terms of recurrence and survival.

The overall aim of this study is to examine different aspects of adjuvant CDK4/i in older early breast cancer patients. In more detail the aims are to investigate the association between geriatric frailty assessment (based on screening by the Geriatric 8 (G8) and Vulnerable Elders Survey-13 (VES-13) screening tools in older breast cancer patients that are to be treated with adjuvant CDK4/6i, and the risk of treatment side effects, discontinuation, patients reported quality of life, and hospitalization. Moreover, the investigators aim at exploring the correlation between frailty as assessed by geriatric screening and dose intensity and this impact on recurrence/survival. As exploratory analysis, different cut-offs for G8 and VES-13 score will be investigated in order to find stronger correlation between vulnerability/frailty and long-term outcomes in this patient cohort, and finally a comparison between the G8 and VES-13 performance.

In detail, the primary objectives are:

1. Association between frailty as assessed by G8 and VES-13 screening and CDK4/6i treatment side effects (adverse event (AE) grade ≥3)
2. Association between frailty as assessed by G8 and VES-13 screening and quality of life after initiating CDK4/6i, as reported by the patient
3. Association between frailty as assessed by G8 and VES-13 screening and hospitalization due to CDK4/6i

   The secondary objectivs are:
4. Association between frailty as assessed by G8 and VES-13 screening and relative dose intensity (RDI, defined as the ratio of the drug dose administered in the actual time, over the planned dose in the planned time) by CDK4/6i and impact on breast cancer recurrence, overall and breast cancer-specific survival after 3, 5 and 10 years, respectively.

As exploratory analysis the following will be performed:

1. Explore whether different cut-offs of G8 and VES-13 score would result in a stronger correlation between vulnerability/frailty and long-term outcomes in this patient cohort. 2. Compare which geriatric screening tool that is more associated to outcomes

ELIGIBILITY:
Inclusion Criteria:

* ≥70 years old
* Female/male
* Completed surgery (primary or after neoadjuvant therapy)
* Starting adjuvant CDK4/6i and endocrine therapy
* Cognitive performance to be able answer questionaries
* No language difficulties

Exclusion Criteria:

* Impaired cognitive function not able to understand the study intention or perform questionaries
* Declining adjuvant CDK4/6i

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: All patients with primary breast cancer, regardless of breast cancer subtype, who are ≥70 years old and starting adjuvant CDK4/6i are included in this trial.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2029-09-01 (Estimated); Study Completion 2039-08-01 (Estimated)

PRIMARY OUTCOMES:
Frailty as assessed by Geriatric 8 (G8) | Baseline
  Geriatric 8 (G8) geriatric screening. 8 questions. Generating total score (0-17). ≤14 indicates frailty.
Frailty as assessed by Vulnerable Elders Survey (VES-13) | Baseline
  Vulnerable Elders Survey (VES-13) geriatric screening, 13 questions. Generating total score (0-10). ≥3 indicates frailty.

SECONDARY OUTCOMES:
Global health status and Quality of Life (QoL) (GHS) | Baseline, 6,12, 24, 36, 60 months from CDK4/6inhibitor initiation.
  Global health status and Quality of Life (QoL) (GHS) comprises the two seven-point Likert scale from the EORTC QLQ-C30 regarding overall health and QoL during the past week.
Summary score | Baseline, 6,12, 24, 36, 60 months from CDK4/6inhibitor initiation
  Comprise all questions from the EORTC QLQ-C30 except for those included in the Global health status and Quality of Life (QoL) (GHS) and a question concerning financial difficulties. Scores range from 0 (no Health-related quality of life (HRQOL)) to 100 (the highest HRQoL).
Ten scales | Baseline, 6,12, 24, 36, 60 months from CDK4/6inhibitor initiation.
  Ten scales include five function scales and five symptom scales from the EORTC-QLQ-C30 and ELD14. Scales included physical, role, and social functioning, fatigue, and pain from the EORTC-QLQ-C30 and maintaining purpose, family support, mobility, future worries, and burden of illness from the EORTC-QLQ ELD14. Scores from all scales range from 0 to 100. High scores for functional scales represent high and healthy functioning, whereas high scores for symptom scales represent high symptomatology.
Adverse events | At 6, 12, 18, 24, 30, 36, 42 months after CDK4/6i initation. Last timepoint is 6 months after ending CDK/6i (e.g 30 months for those treated Abemaciclib and 42 months for those treated with Ribociclib, respectively).
  ≥ Grad 3 adverse events (AE) from CDK4/6 inhibitor (CDK4/6i) according to the CTCAE 5.0
Hospitalization | At 6, 12, 18, 24, 30, 36, 42 months after CDK4/6inhibitor (CDK4/6i) initation. Last timepoint is 6 months after ending CDK/6i (e.g 30 months for those treated Abemaciclib and 42 months for those treated with Ribociclib, respectively).
  Hospitalization rate
Dose adjustment | At 6, 12, 18, 24, 30, 36, 42 months after CDK4/6i initation. Last timepoint is 6 months after ending CDK/6i (e.g 30 months for those treated Abemaciclib and 42 months for those treated with Ribociclib, respectively).
  Change in CDK4/6 inhibitor (CDK4/6i) dosage
Treatment discontinuation | At 6, 12, 18, 24, 30, 36, 42 months after CDK4/6i initation. Last timepoint is 6 months after ending CDK/6i (e.g 30 months for those treated Abemaciclib and 42 months for those treated with Ribociclib, respectively).
  End of CDK4/6inhibitor (CDK4/6i) treatment
Relative dose intensity (RDI) | At 24 and 36 months for those treated with Abemaciclib and Ribociclib, respectively
  RDI; defined as the ratio of the drug dose administered in the actual time, over the planned dose in the planned time
Berast cancer recurrence | At 3, 5, 10 years
  Recurrence (locoregional, distant, in situ)
Survival | At 3, 5, 10 years
  Breast cancer specific and overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Christine Lundgren, MD, Study Chair — Department of Oncology, Jönköping, Region Jönköping County, Jönköping; Sweden,
Locations (6):
- Sweden (6):
  - Department of Oncology, Gävle
  - Department of Oncology, Gothenburg
  - Department of Oncology, Jönköping
  - Department of Oncology, Kalmar
  - Department of Oncology, Linköping
  - Department of Oncology, Örebro

IPD SHARING:
Plan to Share IPD: Undecided